CLINICAL TRIAL: NCT04140110
Title: Second Enhanced Control of Hypertension and Thrombectomy Stroke Study (ENCHANTED2)
Acronym: ENCHANTED2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data Safety Monitoring Board recommendation based on consistent safety concerns that recruitment be discontinued and the data analysed and reported. Protocol amendment planned.
Sponsor: The George Institute for Global Health, China (Other)
Collaborators: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Craig Anderson, Executive Director, The George Institute for Global Health, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENCHANTED2
Record Dates: First submitted 2019-10-22; First posted 2019-10-25 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Large vessel occlusion; Mechanical thrombectomy; Blood pressure management; Antiplatelet therapy; Anticoagulation therapy; Randomised clinical trial
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Different intensities of blood pressure management using locally available intravenous antihypertensive agents
Who Masked: Outcomes Assessor
Masking Description: Open intervention; outcome assessments undertaken by trained research staff who are kept blind to treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Achieving SBP level of <120 mmHg within 1 hour after randomisation, and maintaining this level at least 72 hours.
  Interventions: Other: Intensive BP lowering
- Control group (No Intervention): Maintaining SBP 140-180mmHg, and BP lowering treatment can be given only when BP level ≥150 mmHg in order to achieve the target of ≥140 mmHg, and maintaining this level at least 72 hours.

INTERVENTIONS:
Other: Intensive BP lowering — The aim is to achieve a systolic BP level of <120mmHg within 1 hour after randomisation and to maintain this BP level for the next 72 hours (or until hospital discharge or death if this should occur earlier).
  Arms: Intervention group

SUMMARY:
ENCHANTED2 is an international, multicenter, prospective, randomised, open, blinded end-point assessed (PROBE) trial, to assess different approaches to manage blood pressure (BP) in acute ischemic stroke (AIS) patients who have undergone mechanical thrombectomy (MT). There are two nested substudies evaluating different approaches to secondary prevention in this high-risk stroke population.

DETAILED DESCRIPTION:
Objectives: To determine the effectiveness of more intensive BP lowering target (<120 mmHg) compared to higher BP management target (140-180mmHg) on functional outcome in patients with successful recanalization post-MT for AIS due to large vessel occlusion (LVO).

Inclusion Criteria:

1. Age ≥18 years;
2. Diagnosis of AIS with LVO confirmed by brain imaging;
3. To receive MT <24 hours after AIS onset according to local guidelines;
4. Successful recanalization (TICI score ≥2b) after MT;
5. Sustained systolic BP ≥140 mmHg (defined as 2 successive readings <10 mins) within 3 hours after recanalization;
6. Provide written informed consent (or approved surrogate).

Exclusion Criteria:

1. Unlikely to potentially benefit from therapy (e.g. advanced dementia) or very high likelihood of death within 24 hours post-MT, judged by responsible treating clinician;
2. Other medical illness that interferes with outcome assessments and follow-up (e.g. known significant pre-stroke disability (mRS scores 3-5), advance cancer and renal failure);
3. Definite indication/contraindication to different intensities of BP lowering treatment;
4. Specific contraindications to any of the BP agents to be used (eg, patients who are hypersensitive (allergic) to any of the ingredients);
5. Patients with aortic isthmus stenosis and arteriovenous shunt (exception: patients with haemodynamically inactive dialysis shunt);
6. Women who are lactating;
7. Currently participating in another trial which would interfere with outcome assessments.

Outcome Measures Primary outcome: functional recovery, defined as a shift (improvement) in scores on the modified Rankin scale (mRS) at 90 days.

Secondary outcomes: any intracranial haemorrhage (ICH), symptomatic intracerebral haemorrhage (sICH), early neurological deterioration, imaging assessment (e.g. infarct size, edema volume), death, disability, HRQoL, duration of hospitalization, residence; and health service use for calculation of resources and costs.

Randomisation and intervention: Randomisation is via a central internet-based system, stratified by site, time from symptom onset to recanalization (<6, ≥6 hours), baseline neurological impairment on the National Institutes for Health Stroke Scale (NIHSS <17 vs ≥17), to ensure balance in key prognostic factors.

Intensive BP lowering group: to commence intravenous BP lowering therapy immediately after randomization, with systolic BP target (<120 mmHg) achieved within 1 hour, and maintained for at least 72 hours (or hospital discharge if earlier).

Control group: to receive guideline-recommended BP control strategy to maintain BP level 140-180 mmHg after MT procedure, but BP lowering treatment given only for BP ≥150 mmHg to achieve target ≥140 mmHg.

Substudies: Patients enrolled in main study can also be randomised into 2 substudies according to separate eligibility criteria. Both are pilot studies embedded in main trial to recruit as many patients to inform sample size estimates for a further main study.

Substudy #1: Timing of anticoagulation Objective: To determine the effectiveness of early initiation of anticoagulation (at Day 4±2 of stroke onset) compared with late initiation (at Day 12±2) on a composite outcome of recurrent AIS, sICH, systemic embolism and/or death within 90 days in patients with AF-related AIS due to LVO who receive MT. Randomisation (allocation 1:1 ratio) via same system as main study and stratified by site and randomisation of BP intervention. Randomised patients will be allocated to either early group of initiating OAC therapy at Day 4±2 day of stroke onset, or late group of initiating OAC therapy at Day 12±2 of stroke onset. Primary outcome: composite of recurrent AIS, sICH, systemic embolism and/or vascular death within 90 days after randomisation.

Substudy #2: Duration of dual antiplatelet therapy (DAPT):

Objective: To determine the effectiveness of short duration of DAPT (<6 weeks) compared with standard duration (3 months or more) on recurrence rate within 12 months in patients with AIS due to large artery atherosclerosis (LAA) who are eligible for DAPT post-MT. Randomisation (allocation 1:1 ratio) will be done via the same system as the main study and stratified by site and randomisation of BP intervention. Randomised patients will be allocated to either short duration group of receiving DAPT (aspirin 100 mg and clopidogrel 75 mg per day) for 6 weeks, or standard duration group receiving DAPT for 3 months. DAPT is started <48 hours post-randomization, and maintained changed to antiplatelet monotherapy (aspirin or clopidogrel) thereafter. Primary outcome is new stroke event (AIS or ICH) over 12 months.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years; Diagnosis of AIS with LVO confirmed by brain imaging; To receive MT <24 hours after AIS onset according to local guidelines; Successful recanalization (TICI score ≥2b) after MT; Sustained systolic BP ≥140 mmHg (defined as 2 successive readings <10 mins) within 3 hours after recanalization; Provide written informed consent (or approved surrogate).

Exclusion Criteria:

Unlikely to potentially benefit from therapy (e.g. advanced dementia) or very high likelihood of death within 24 hours post-MT, judged by responsible treating clinician; Other medical illness that interferes with outcome assessments and follow-up (e.g. known significant pre-stroke disability (mRS scores 3-5), advance cancer and renal failure); Definite indication/contraindication to different intensities of BP lowering treatment; Specific contraindications to any of the BP agents to be used (eg, patients who are hypersensitive (allergic) to any of the ingredients); Patients with aortic isthmus stenosis and arteriovenous shunt (exception: patients with haemodynamically inactive dialysis shunt); Women who are lactating; Currently participating in another trial which would interfere with outcome assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 816 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Level of disability | 90 days (3 months)
  a shift (improvement) in scores (0-6) on the modified Rankin scale

SECONDARY OUTCOMES:
intracerebral hemorrhage (ICH) | 90 days
  any or symptomatic ICH (sICH) after MT
Imaging endpoints | 24-48 hours
  infarct size growth
Imaging endpoints | Day 7
  edema volume
Death or neurological severity | 7 days
  Death or dependency measured by National Institutes of Health stroke scale (NIHSS)
Others | 90 days
  Death or major disability (mRS 3-6); separately on death and disability (mRS 3-5); health-related quality of life (HRQoL) using EQ-5D; duration of hospitalisation; residence and hospital service cost.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Anderson, Principal Investigator — The George Institute for Global Health, China; Jianmin Liu, Principal Investigator — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with bona fide researchers after after publication of the main results, based on a submitted protocol to the research office of The George Institute for Global Health, Sydney Australia.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data sharing will be available from 12 months after publication of the main results.
Access Criteria: 1. The data sharing will be only for the purposes of health and medical research and within the constraints of the consent under which the data were originally gathered.
  2. The Custodian of the Collection will not consider any Proposals for data sharing that unblind, or potentially unblind, randomised comparisons in active / ongoing trials.
  3. Requesters should be employees of a recognised academic institution, health service organisation, commercial research organisation or from the pharmaceutical industry. Requesters must have experience in medical research.
  4. Requesters must be able to demonstrate through their peer review publications in the area of interest their ability to carry out the proposed use of the requested dataset from a Collection.
  5. The Requesters must not have a conflict of interest that may potentially influence their interpretation of any analyses.
URL: http://georgeinstitute.org.au

REFERENCES:
- [Derived] Zhang X, Ren X, Zhang Y, Zhang Y, Zhang L, Shen H, Li Z, Xing P, Zhang P, Hua W, Shen F, Tian B, Chen W, Han H, Zhang L, Xu C, Li T, Gao Y, Zhou Y, Zuo Q, Dai D, Zhao R, Li Q, Huang Q, Xu Y, Chen X, Li Q, Song L, Anderson CS, Yang P, Liu J; ENCHANTED2/MT Collaboration. Interaction of brain imaging features and effects of intensive blood pressure lowering after endovascular treatment for acute ischaemic stroke: the pre-specified secondary analyses of ENCHANTED2/MT trial. EClinicalMedicine. 2025 Apr 21;83:103197. doi: 10.1016/j.eclinm.2025.103197. eCollection 2025 May. PMID 40330548
- [Derived] Yang P, Song L, Zhang Y, Zhang X, Chen X, Li Y, Sun L, Wan Y, Billot L, Li Q, Ren X, Shen H, Zhang L, Li Z, Xing P, Zhang Y, Zhang P, Hua W, Shen F, Zhou Y, Tian B, Chen W, Han H, Zhang L, Xu C, Li T, Peng Y, Yue X, Chen S, Wen C, Wan S, Yin C, Wei M, Shu H, Nan G, Liu S, Liu W, Cai Y, Sui Y, Chen M, Zhou Y, Zuo Q, Dai D, Zhao R, Li Q, Huang Q, Xu Y, Deng B, Wu T, Lu J, Wang X, Parsons MW, Butcher K, Campbell B, Robinson TG, Goyal M, Dippel D, Roos Y, Majoie C, Wang L, Wang Y, Liu J, Anderson CS; ENCHANTED2/MT Investigators. Intensive blood pressure control after endovascular thrombectomy for acute ischaemic stroke (ENCHANTED2/MT): a multicentre, open-label, blinded-endpoint, randomised controlled trial. Lancet. 2022 Nov 5;400(10363):1585-1596. doi: 10.1016/S0140-6736(22)01882-7. Epub 2022 Oct 28. PMID 36341753
- [Derived] Song L, Yang P, Zhang Y, Zhang X, Chen X, Li Y, Shen H, Zhang L, Li Z, Zhang Y, Xing P, Zhang P, Zhou Y, Ren X, Billot L, Wang X, Parsons MW, Butcher K, Campbell B, Robinson T, Goyal M, Dippel D, Roos Y, Majoie C, Liu J, Anderson CS; for ENCHANTED-MT Investigators. The second randomized controlled ENhanced Control of Hypertension ANd Thrombectomy strokE stuDy (ENCHANTED2): Protocol and progress. Int J Stroke. 2023 Mar;18(3):364-369. doi: 10.1177/17474930221120345. Epub 2022 Aug 24. PMID 35924814

DOCUMENTS (2):
  • Study Protocol (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT04140110/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT04140110/SAP_001.pdf